CLINICAL TRIAL: NCT01832831
Title: Anatomical and Functional Differences Between Continent and Incontinent Men Post Radical Prostatectomy
Status: Terminated | Type: Observational
Why Stopped: The study was completed as planned
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Anne Pelletier-Cameron, Associate Professor, Urology, University of Michigan
Other Study IDs: HUM00035833
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer; Post Prostatectomy Incontinence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Continent Men
- Incontinent Men

SUMMARY:
One out of every six men will be diagnosed with prostate cancer and post prostatectomy up to 75% report urinary incontinence. There are many hypotheses about the exact cause of post prostatectomy stress incontinence (PPI). Existing studies have focused on surgical or cadaveric dissections to define structures responsible for PPI. Contemporary 3T MRI now allows three dimensional, sub-millimeter resolution of the human pelvis and clearly demonstrates pelvic anatomy without the distortion of dissection. It is our overarching hypothesis that PPI is multifactorial and occurs because of a combination of specific anatomical and functional impairments. We propose conducting a case control study with matching for age and race to compare the MRI anatomy and urinary tract function on urodynamics between 20 men with PPI (cases) and 20 men who are continent post prostatectomy (controls) who are all a minimum of 12 months post surgery. We will use static and dynamic MRI at 3 Tesla to make objective measurements of the bladder neck, external urethral sphincter, pelvic floor, urethral anastomotic fibrosis, and urethral hypermobility- all believed to play a large part in continence. Multi-channel urodynamic studies will also be performed to assess the leak point and maximum urethral closure pressure. All cases and controls will complete standardized questionnaires - the AUA symptom index and the Incontinence Severity Index as a quality of life measure. This study is needed to provide critical information about causes of male PPI, a quality of life altering voiding dysfunction, and will assist with the advancement of pharmacological and surgical treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Only men will be included since this is a study of post prostatectomy incontinence. Cases will be comprised of men who are post radical retropubic or laparoscopic (robotic) prostatectomy who have stress urinary incontinence based on history and a minimum of 50 grams of urine loss on 24 hour pad weights. Controls will be comprised of men who are post radical retropubic or laparoscopic (robotic) prostatectomy who do not have any kind or amount of incontinence based on history. Cases and controls will be matched for both age and race these have been shown to alter anatomical appearance of structures and lower urinary tract function.

Exclusion Criteria:

* Criteria for both groups include urge incontinence, urinary retention, neurologic disease, insulin dependent diabetes, high dose steroid use, pre-surgical abnormal voiding function or incontinence, prior pelvic radiation or urologic surgery, any prior incontinence surgery, current medical therapy for incontinence or a perineal route of radical prostatectomy since this had been shown to give a distinctly different appearance on MRI compared to the laparoscopic or retropubic approach. Any patient with pelvic or systemic recurrence of their prostate cancer will also be excluded. Any man with relative or absolute contraindications to MRI such as implants or claustrophobia will be excluded.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Thickness and length of both the smooth muscle and striated muscle external urethral sphincter | 2 years
  Structural assessment
Posterior urethral length from the bladder neck to the perineal membrane. | 2 years
  Structural assessment
Levator ani thickness | 3 years
  Structural assessment
Thickness and length of anastomotic fibrosis in both sagittal and axial planes | 3 years
  Structural assessment
Maximal urethral closure pressure | 3 years
  Functional assessment
Increase in urethral pressure during maximal muscle contraction | 3 years
  Functional assessment
Urethral hypermobility on MRI | 3 years
  Functional assessment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Pelletier-Cameron, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan